CLINICAL TRIAL: NCT04506112
Title: Optimizing Cardiac Rehabilitation by Integrating Sleep Therapeutics
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator leaving institution. Aim 3 was not initiated.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E3393-W; RX003393 (Registry Identifier: Department of Veterans Affairs)
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Sleep Wake Disorders; Sleep Disturbance; Sleep-Related Impairment
Keywords: Veterans; Cardiac Rehabilitation
MeSH Terms: conditions — Sleep Wake Disorders; Parasomnias | interventions — Acclimatization; Cardiac Rehabilitation

STUDY DESIGN:
Intervention Model Description: Pilot randomized trial with participants assigned to one of two groups in parallel for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TranS-C + Usual Care (Experimental): Participants in this group will receive TranS-C and will continue with care in cardiac rehabilitation as usual.
  Interventions: Behavioral: Transdiagnostic Sleep and Circadian Intervention (TranS-C), adapted for cardiac rehabilitation
- Usual Care (No Intervention): Participants in this group will receive only usual care and thus will continue with care in cardiac rehabilitation as usual.

INTERVENTIONS:
Behavioral: Transdiagnostic Sleep and Circadian Intervention (TranS-C), adapted for cardiac rehabilitation — Participants will complete the TranS-C intervention as adapted for cardiac rehabilitation. TranS-C is a behavioral intervention that is rooted in basic sleep and circadian science and draws from empirically-supported treatments including Cognitive Behavioral Therapy for Insomnia (CBT-I), Interpersonal and Social Rhythm Therapy (IPSRT), chronotherapy, and light therapy. It was designed to promote sleep health across a range of sleep problems. Participants in this group will also continue to receive care as usual, cardiac/sleep-related or otherwise.
  Other Names: TranS-C
  Arms: TranS-C + Usual Care

SUMMARY:
The study aims are to: 1) optimize the Transdiagnostic Sleep and Circadian Intervention (TranS-C) for delivery to Veterans in cardiac rehabilitation, 2) test and refine the adapted TranS-C treatment manual and protocol, and 3) conduct a pilot randomized trial to establish the feasibility, acceptability, and plausibility of the intervention protocol and study procedures.

DETAILED DESCRIPTION:
Aim 1 will involve formative work to optimize the TranS-C manual and protocol for delivery in Cardiac Rehabilitation, with input from Veterans and provider stakeholders. Aim 2 will involve a preliminary test and refinement of the adapted TranS-C manual and protocol with a small sample of Veterans who are participating in cardiac rehabilitation and report sleep disturbance and/or sleep-related impairment. Aim 3 will involve a pilot randomized trial to establish the feasibility, acceptability, and plausibility of the intervention protocol and study procedures. Veterans in cardiac rehabilitation with sleep disturbance and/or sleep-related impairment will be randomized to TranS-C + Usual Care or Usual Care. Treatment satisfaction will be assessed at 3-months; sleep disturbance and sleep-related impairment, disability and functioning, and health-related quality of life will be assessed at baseline, 3-months, and 6-months to determine measure responsiveness and provide preliminary insight into treatment effects.

Of note, information provided in this entry (e.g., design, eligibility criteria, outcomes, etc.) pertains only to Aim 3 which includes the pilot randomized trial. Consistent with Stage I of the NIH stage model of behavioral intervention development research, results from Aim 1 and 2 activities may lead to modifications to the pilot protocol and procedures in Aim 3.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Age 18 years or older
* Referred for VAPHS cardiac rehabilitation
* Self-reported sleep disturbance or sleep-related impairment, determined by PROMIS Sleep Disturbance T-score at least 55 (raw score at least 25) or PROMIS Sleep-Related Impairment T-score at least 55 (raw score at least 20)
* English language fluency
* Willing and able to voluntarily participate in a behavioral sleep intervention clinical research study
* Willing to permit study personnel access to VA EHR
* Willing to permit study personnel to communicate with routine VA healthcare providers
* Willing and able to participate in outpatient cardiac rehabilitation at VAPHS

Exclusion Criteria:

* Moderate to severe cognitive impairment
* Active suicidal ideation, plan, or intent
* Current moderate to severe alcohol or substance use disorder
* Current severe symptoms of depression, anxiety, mania/hypomania, psychosis, or PTSD
* Currently engaged in a non-pharmacological intervention for sleep
* Currently working night shifts
* Currently pregnant and/or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-04-16 (Actual); Study Completion 2023-04-16 (Actual)

PRIMARY OUTCOMES:
Multidimensional Treatment Satisfaction Measure | 3 months
  Self-report measure of patient satisfaction with behavioral intervention process and outcomes. Subscale scores range from 0-4. Higher scores are suggestive of greater satisfaction with treatment.
Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v 1.0-Sleep Disturbance 8a from Baseline to 3 and 6 months | Baseline to 3 and 6 months
  Validated self-report measure of global sleep disturbance over the preceding 7 days. Produces raw score and T-score values, where 50 is the mean of the reference population and 10 is the standard deviation.
  Higher scores are indicative of greater sleep disturbance.
Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v 1.0-Sleep Related Impairment 8a from Baseline to 3 and 6 months | Baseline to 3 and 6 months
  Validated self-report measure of sleep-related impairment over the preceding 7 days. Produces raw score and T-score values, where 50 is the mean of the reference population and 10 is the standard deviation. Higher scores are indicative of greater sleep-related impairment.
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) from Baseline to 3 and 6 months | Baseline to 3 and 6 months
  Validated self-report measure of disability and functioning associated with physical and mental disorders. The WHODAS 2.0 contains 36-items that assess functioning in the domains of cognition, mobility, self-care, getting along, life activities, and participation over the preceding 30 days. The outcome of interest is the WHODAS 2.0 summary score. Using the complex scoring method, scores range from 0 to 100. Higher scores are indicative of greater disability.
MacNew Heart Disease Health-Related Quality of Life Questionnaire (MacNew) from Baseline to 3 and 6 months | Baseline to 3 months and 6 months
  Validated self-report measure of health-related quality of life in patients with heart disease. Contains 27 items that assess physical limitations, emotional function, social function, and symptoms common in heart disease (e.g., angina/chest pain, shortness of breath, fatigue, aching legs). The outcome of interest is the total health-related quality of life score. Scores range from 1 to 7. Higher scores are indicative of higher levels of health-related quality of life.

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) from Baseline to 3 and 6 months | Baseline to 3 and 6 months
  Validated performance-based measure of physical function. Includes assessments of gait speed, functional strength, and standing balance. Total scores range from 0 to 12. Higher scores are indicative of better performance.
Physical Performance Test (PPT)from Baseline to 3 and 6 months | Baseline to 3 and 6 months
  Validated performance-based measure of physical functioning. Requires participants to perform 7 activities that simulate activities of daily living (e.g., writing a sentence, putting on a jacket). Scores range from 0 to 28. Higher scores are indicative of better performance.
Life Space Assessment from Baseline to 3 and 6 months | Baseline to 3 and 6 months
  Validated self-report measure of life space mobility (i.e., the spatial area in which a person navigates). Respondents indicate how far and how often they have traveled to various places (e.g., in immediate neighborhood, outside immediate town or community) in the past 4 weeks. Composite scores range from 0 to 120. Higher scores are suggestive of greater life space mobility.
World Health Organization Quality of Life-BREF (WHOQOL-BREF) from Baseline to 3 and 6 months | Baseline to 3 and 6 months
  Validated self-report measure of quality of life. Contains 26 items that assess and yield scores representative of quality of life in the domains of physical health, psychological health, social relationships, and environment. Domain scores range from 0 to 100. Higher scores are indicative of higher quality of life.

OTHER OUTCOMES:
Pittsburgh Sleep Quality Index from Baseline to 3 and 6 months | Baseline to 3 and 6 months
  Validated self-report measure of global sleep quality. Items assess past-month subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medication, and daytime dysfunction. Global sleep quality scores range from 0 to 21. Higher scores are indicative of worse sleep quality.
Insomnia Severity Index from Baseline to 3 and 6 months | Baseline to 3 and 6 months
  Validated self-report measure of insomnia symptoms over the past 2 weeks. Contains 7 items assessing severity of insomnia symptoms. Scores range from 0 to 28. Higher scores are indicative of greater insomnia severity.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlan A. Tighe, PhD MA, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Final data sets underlying publications resulting from the proposed research may be shared.
Time Frame: Prior to the end of the study.
Access Criteria: A Limited Dataset (LDS) may be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.